CLINICAL TRIAL: NCT04431921
Title: Assessment of Functional Capacity, Pain, Cognitive and Respiratory Functions in Lung Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Kılıç, Physiotherapist, Hacettepe University
Other Study IDs: GO17/555
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Lung Neoplasm; Survivorship
Keywords: Respiratory muscles; Pain; Cognitive dysfunction
MeSH Terms: conditions — Lung Neoplasms; Pain; Cognitive Dysfunction | interventions — Functional Residual Capacity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung cancer patients: Lung cancer survivors who had stable conditions and routine follow-up at Hacettepe University Oncology Hospital
  Interventions: Diagnostic Test: Functional capacity
- Healthy subjects: No health problems related or affect outcome measure parameters examined in this study.
  Interventions: Diagnostic Test: Functional capacity

INTERVENTIONS:
Diagnostic Test: Functional capacity — Six minute walk test used assessment of functional capacity. For respiratory function mouth pressures, for cognitive functions MoCA scale and for pain assessment pain threshold and tolerance test assessed.
  Other Names: Exercise capacity

SUMMARY:
Serious side effects occurs with disease and treatments in survival after lung cancer. For this reason, functional capacity, cognitive status, pain perception and respiratory functions may be affected in lung cancer. The purpose of this study was to evaluate respiratory function, respiratory muscle strength and endurance, functional capacity, pain, cognitive status level, and physical activity in lung cancer patients and compare with the findings of healthy subjects

DETAILED DESCRIPTION:
This study was participated lung cancer patients survivors. Patients' pulmonary function test, functional capacity, respiratory muscle strength and endurance, pain and cognitive status was assessed and recorded.

Pulmonary function testing (PFT), mouth pressure measurement (MIP- maximal inspiratory pressure and MEP- maximal expiratory pressure), respiratory muscle endurance test, six minute walk test (6MWT) and pain threshold and tolerance test were used. In addition to physiological measurements, the Montreal Cognitive Assessment (MoCA) scale was used to evaluate cognitive status, the International Physical Activity Questionnaire (IPAQ) was used to determine the level of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Cooperation
* lung cancer patients who had a stable condition

Exclusion Criteria:

* Active cancer treatments
* Brain metastasis story
* Any orthopedic disease impairs walking, balance

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients -> patients who were not under active cancer treatments Healthy -> No lung disease and systemic disease that affected outcome measure
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Functional capacity | 15 minutes
  Six minute walk test: Distance walked in six minute was recorded

SECONDARY OUTCOMES:
Respiratory muscle strength assessment | 10 minutes
  Respiratory muscle strength was evaluated by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP).
Respiratory muscle endurance | 10 minutes
  Pressure time unit: A constant load test was used to evaluate respiratory muscle endurance. Using a PowerBreathe device (HaB International Ltd., Southam, UK), the participants were asked to breathe maintaining a constant threshold (60% of MIP) until task failure, and the test duration was recorded. Results were obtained by multiplying the set pressure by the test duration
Pulmonary functions test | 15 minutes
  pulmonary functions assessment via spirometry
Cognition using MoCA-Test | 10 minutes
  Cognitive function was evaluated with the secreening tool the Montreal Cognitive Assessment (MoCA). The MoCA is a 30-point screening tool. Higher scores mean a better outcome.
Pressure pain threshold assessment | 15 minute
  Pressure pain threshold was evaluated via algometer. The pressure at which the individual first reported pain was recorded.
Pressure pain tolerance assessment | 15 minute
  Pressure pain tolerance test was evaluated via algometer.The pressure at which the individual last pressure point at which they could endure the pain was recorded.
Physical activity level | 5 minutes
  International Physical Activity Questionnaire-Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Deniz Inal-Ince, Professor, Study Chair — Hacettepe University; Melda Saglam, PhD, Study Chair — Hacettepe University; Ebru Calik-Kütükcü, PhD, Study Chair — Hacettepe University; Hulya Arikan, Professor, Study Chair — Hacettepe University; Saadettin Kilickap, Professor, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided